CLINICAL TRIAL: NCT03656640
Title: A Prospective, Multicenter Observational Trial Assessing the Safety and Efficacy of Gammanorm® in Autoimmune Diseases
Brief Title: Trial Assessing Safety and Efficacy of Gammanorm® in Autoimmune Diseases
Status: Terminated | Type: Observational
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Other Study IDs: IMMUNORM
Record Dates: First submitted 2017-11-30; First posted 2018-09-04 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Receiving Gammanorm®: Patients Receiving Gammanorm®
  Interventions: Drug: Gammanorm

INTERVENTIONS:
Drug: Gammanorm — Patients already receiving Gammanorm will be observed over the course of 2 years every 3 months. Gammanorm will be given standard of care.

SUMMARY:
This observational trial assesses the safety and efficacy of Gammanorm® in autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Adult man or woman older than 18 years,
2. Patient with autoimmune disease such as CIDP, MMN, PM, DM, MI, ITP, NAM or any other off-label use of Gammanorm®,
3. Patient who has a prescription of Gammanorm® treatment for immunomodulation,
4. Patient accepting to participate in the study by oral consent after having received oral and written information on the study.

Exclusion Criteria:

1. Patient treated with Gammanorm® for immune substitution, or other authorized use
2. Patient who refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men and women over 18 prescribed Gammanorm with autoimmune disease or any other off-label use of Gammanorm who are willing to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of Gammanorm® in terms of adverse event rate in patients receiving the off-label treatment in immunomodulation. | 24 months
  Evaluate the safety of Gammanorm® in terms of adverse event rate in patients receiving the off-label treatment in immunomodulation.

SECONDARY OUTCOMES:
SMOG score | 24 months
  For patients with idiopathic thrombocytopenic purpura, efficacy will be assessed using the SMOG score. SMOG score : Bleeding manifestations are grouped into three major domains: skin (S), visible mucosae (M), and organs (O), with gradation of severity (SMOG). Each bleeding manifestation is assessed at the time of examination. Severity is graded from 0 to 3 or 4, with grade 5 for any fatal bleeding.
Rankin score | 24 months
  For patients with Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal motor neuropathy (MMN), efficacy will be assessed using the Rankin score
MRC | 24 months
  For patients with Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal motor neuropathy (MMN), efficacy will be assessed using the MRC. MRC (Medical research council) scale for testing muscle : The muscle scale grades muscle power on a scale of 0 to 5 in relation to the maximum expected for that muscle (5= Normal power , 0= No contraction visible or palpable).
ONLS | 24 months
  For patients with Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) and Multifocal motor neuropathy (MMN), efficacy will be assessed using the ONLS (overall neuropathy limitations score). Score ONLS (Overall Neuropathy Limitation Scale) : The OLNS focuses on upper and lower limb functions, and consists of a checklist for interviewing patients. It is scored from 0 to 5 on the upper limb section and from 0 to 7 on the lower limb section. A score of 0 indicates no limitations (the ceiling of the scale) and a score of 5 or 7 indicates no purposeful movement.
Muscular Testings and Myositis Functional Rating Scale | 24 months
  For patients with inflammatory myopathies including dermatomyositis (DM), polymyositis (PM), inclusion body myositis (IBM), and autoimmune necrotizing myopathy (AINM), efficacy will be assessed using the muscular testings and myositis functional rating scale
Evaluate treatment compliance | 24 months
  Evaluate treatment compliance in terms of number of infusions per week
Evaluate reasons for stopping the treatment | 24 months
  Evaluate reasons for stopping the treatment by categorizing across the study the reasons subjects stopped treatment.
Patient satisfaction regarding Gammanorm | 24 months
  Evaluate patient satisfaction with use of patient diaries where the patient will complete a questionnaire on Life Quality Index (LQI)
Patient Quality of Life regarding Gammanorm | 24 months
  Evaluate patient quality of life with use of patient diaries where the patient will complete a questionnaire on quality of life (SF-12)

CONTACTS AND LOCATIONS:
Locations (3):
- France (2):
  - APHP - Pitie Salpetriere, Paris
  - Chu de Rouen - Bois Guillaume, Rouen
- CHU de la Martinique- Hopital Pierre Zobda Quitman, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: Undecided